CLINICAL TRIAL: NCT02831933
Title: ENSIGN: Phase II Window of Opportunity Trial of Stereotactic Body Radiation Therapy and In Situ Gene Therapy Followed by Nivolumab in Metastatic Squamous or Non-Squamous Non-Small Cell Lung Carcinoma and Metastatic Uveal Melanoma
Brief Title: Trial of Radiation and Gene Therapy Before Nivolumab for Metastatic Non-Small Cell Lung Carcinoma and Uveal Melanoma
Acronym: ENSIGN
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Eric Bernicker, MD (Other)
Responsible Party: Sponsor-Investigator, Eric Bernicker, MD, Sponsor-Investigator/Principal Investigator, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00014976
Record Dates: First submitted 2016-07-01; First posted 2016-07-13 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Lung Squamous Cell Carcinoma Stage IV; Nonsquamous Nonsmall Cell Neoplasm of Lung; Metastatic Uveal Melanoma
Keywords: lung cancer; metastatic; gene therapy; immunotherapy; melanoma; uveal
MeSH Terms: conditions — Uveal Melanoma; Lung Neoplasms; Neoplasm Metastasis; Melanoma | interventions — Valacyclovir; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): ADV/HSV-tk (5 x 1011 viral particles) in a 2-mL total volume will be injected intratumorally on day 0 of the study.
  Valacyclovir will be orally administered at a dose of 2 g three times daily for 14 days. Valacyclovir treatment will be administered 24 hours after the gene vector injection from day 1 to day 15 of the study.
  SBRT of 30 gray (Gy; 6 Gy X 5 fractions) will be administered over 2 weeks from day 2 to day 16 of the study.
  Nivolumab (480 mg) will be administered intravenously over 30 minutes every 4 weeks starting on day 17 of the study and continuing until disease progression, unacceptable toxicity, or up to 12 months in patients without disease progression.
  Interventions: Biological: ADV/HSV-tk; Drug: Valacyclovir; Radiation: SBRT; Drug: nivolumab

INTERVENTIONS:
Biological: ADV/HSV-tk — Replication-defective recombinant adenovirus vector
Drug: Valacyclovir — Prodrug of the antiviral drug acyclovir
  Other Names: valacyclovir hydrochloride
Radiation: SBRT — Low-dose SBRT
Drug: nivolumab — Fully human immunoglobulin (Ig) G4 anti-PD-1 monoclonal antibody
  Other Names: Opdivo

SUMMARY:
This is a Phase II trial to determine the efficacy and safety of in situ gene therapy and stereotactic body radiation therapy (SBRT) used as a window of opportunity treatment before nivolumab in patients with metastatic squamous or non-squamous non-small cell lung carcinoma (NSCLC) and metastatic uveal melanoma. In situ gene therapy will consist of adenovirus-mediated expression of herpes simplex virus thymidine kinase (ADV/HSV-tk) plus Valacyclovir therapy.

DETAILED DESCRIPTION:
This is a Phase II trial to determine the efficacy and safety of in situ gene therapy and stereotactic body radiation therapy (SBRT) used as a window of opportunity treatment before nivolumab in patients with metastatic squamous or non-squamous non-small cell lung carcinoma (NSCLC) and metastatic uveal melanoma. In situ gene therapy will consist of adenovirus-mediated expression of herpes simplex virus thymidine kinase (ADV/HSV-tk) plus Valacyclovir therapy. Male or female patients aged ≥18 years with histologically or cytologically confirmed metastatic squamous or non-squamous NSCLC whose disease has progressed after a platinum-based chemotherapy and a single-agent immunotherapy OR histologically or cytologically confirmed metastatic uveal melanoma that is immunotherapy naive are eligible to participate in the study. NSCLC patients with EGFR or ALK genomic tumor aberrations are eligible only if they have had disease progression on FDA-approved therapy for these aberrations. ADV/HSV-tk (5 x 1011 viral particles) in a 2-mL total volume will be injected intratumorally on day 0 of the study. Valacyclovir will be orally administered at a dose of 2 g three times daily for 14 days. Valacyclovir treatment will be administered 24 hours after the gene vector injection from day 1 to day 15 of the study. SBRT of 30 gray (Gy; 6 Gy X 5 fractions) will be administered over 2 weeks from day 2 to day 16 of the study. Nivolumab (480 mg) will be administered intravenously over 30 minutes every 4 weeks starting on day 17 of the study and continuing until disease progression, unacceptable toxicity, or up to 12 months in patients without disease progression. The primary endpoint will be the objective response rate (ORR) of ADV/HSV-tk + Valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before nivolumab in patients with metastatic squamous or non-squamous NSCLC. Both RECIST 1.1 and modified immune-related response criteria (irRC; derived from RECIST 1.1) will be used to assess treatment response. Secondary endpoints will include a) clinical benefit rate (CBR); b) duration of response (DoR); c) overall survival (OS) and progression-free survival (PFS) rates; d) safety and toxicity (toxicity will be defined as any treatment-related death or any ≥ grade 3 toxicity excluding alopecia and constitutional symptoms as assessed by the NCI CTCAE v4.03); and e) immune-mediated antitumor activity (assessed by RECIST 1.1 and modified irRC) of ADV/HSV-tk plus Valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before nivolumab.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age.
* Histologically or cytologically confirmed stage IV, metastatic squamous or non-squamous NSCLC that has progressed after a platinum-based chemotherapy and after a single-agent immunotherapy OR histologically or cytologically confirmed metastatic uveal melanoma that is immunotherapy naive
* Evaluable or measurable disease as per RECIST 1:1, a target lesion of suitable diameter (at least 5 mm) for SBRT, and a non-target lesion of at least 1 cm in diameter for abscopal effect evaluation.
* ≥ 4 weeks since any major surgery.
* A 2-week washout period post any prior systemic anticancer therapy, RT, and/or investigational therapy is required prior to trial entry. Subject should be adequately recovered from the acute toxicities of any prior therapy.
* Life expectancy greater than or equal to 6 months.
* Eastern Cooperative Oncology Group performance status of 0-1.
* Adequate bone marrow function:

  * Absolute neutrophil count ≥ 1.5 x 10^9/L (without granulocyte colony stimulating factor support within 2 weeks of laboratory test used to determine eligibility)
  * Platelets ≥ 100 x 10^9/L (without transfusion within 2 weeks of laboratory test used to determine eligibility)
  * Hemoglobin ≥ 8 g/dL (without blood transfusion)
  * White blood cell count > 2,500/uL and < 15,000/uL
  * Lymphocyte count ≥ 500/uL
* Adequate liver function (NSLC Cohort):

  * Serum bilirubin less than or equal to 1.0 X upper limit of normal (ULN; patients with known Gilbert's disease who have serum bilirubin level less than or equal to 3 X ULN may be enrolled)
  * Serum transaminases (aspartate transaminase [AST] or alanine transaminase [ALT]) activity less than or equal to 2.5 X ULN with normal alkaline phosphatase (patients with liver metastases less than or equal to 5 x ULN) OR AST and ALT less than or equal to 1.5 X ULN with an alkaline phosphatase greater than 2.5 X ULN
* Adequate liver function (uveal melanoma cohort):

  * Serum bilirubin less than 1.5 ULN (patients with known Gilbert's disease who have serum bilirubin level 3 ULN may be enrolled)
  * Serum transaminases (AST or ALT) activity less than or equal to 4 ULN with normal alkaline phosphatase (patients with liver metastases less than or equal to 5 x ULN) OR AST and ALT less than or equal to 1.5 ULN with an alkaline phosphatase greater than or equal to 2.5 ULN
* International normalized ratio and activated partial thromboplastin time (aPTT) less than or equal to 1.5 X ULN (unless patient is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants)
* Adequate renal function: serum creatinine less than 2 X ULN.
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 7 days prior to the administration of the first study treatment. Women must not be lactating.
* WOCBP and men must practice an effective method of birth control
* Signed informed consent to participate in the study must be obtained from patients after they have been fully informed of the nature and potential risks of the study by the investigator (or his/her designee) with the aid of written information.
* Willing to provide biopsies as required by the study.

Exclusion Criteria:

* Prior treatment with gene therapy.
* Any immunotherapy within 2 weeks of study treatment start (NSCLC cohort only).
* Prior treatment with immunotherapy (uveal melanoma cohort only)
* Patients with EGFR or ALK genomic tumor aberrations that have not received any FDA-approved therapy for these aberrations (NSCLC cohort only).
* Oxygen-dependent chronic obstructive pulmonary disease (NSCLC cohort only).
* Patients requiring oral prednisone for emphysema management (NSCLC cohort only).
* History of liver disease, such as cirrhosis or active/chronic hepatitis B or C.
* History of or current alcohol misuse/abuse within the past 12 months.
* Known gallbladder or bile duct disease (i.e., infection or cholecystitis) or acute or chronic pancreatitis.
* Major surgery within 4 weeks prior to study enrollment.
* Uncontrolled brain or leptomeningeal metastases or brain or leptomeningeal metastases requiring continued glucocorticoid treatment. Patients who have been treated at least 4 weeks prior to enrollment and have a CT or magnetic resonance imaging scan of the brain showing no evidence of disease progression within 4 weeks of enrollment are eligible.
* Congestive heart failure: New York Heart Association class III or IV heart failure or unstable angina.
* History of syncope or family history of idiopathic sudden death.
* Sustained or clinically significant cardiac arrhythmias including sustained ventricular tachycardia, ventricular fibrillation, clinically significant bradycardia, advanced heart block (Mobitz II or higher atrioventricular nodal block), prolonged heart rate-corrected QT interval (longer than 470 milliseconds), or history of acute myocardial infarction. (The QT interval is the time between the start of the Q wave and the end of the T wave in the cardiac electrical cycle)
* Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes or Parkinson's disease), human immunodeficiency virus (HIV), cirrhosis, uncontrolled hypothyroidism, or cardiac failure.
* Presence of active or suspected acute or chronic uncontrolled infection or history of immunocompromise, including a positive HIV test result.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect patient participation in the study such as severely impaired lung function, any active (acute or chronic) or uncontrolled infection/disorders, and nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the study therapy.
* Known or suspected allergy or hypersensitivity to any component of nivolumab or its analogues or any component of the proposed regimen (gene vector/Valacyclovir).
* Inability to swallow food or any condition of the upper gastrointestinal tract that precludes administration of oral medications (Valacyclovir).
* Any active malignancy except for non-melanoma skin cancer or in situ cervical cancer or treated cancer from which the patient has been continuously disease free for more than 5 years.
* Pregnant or breastfeeding women or women/men able to conceive and unwilling to practice an effective method of birth control.
* Unwilling or unable to comply with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2020-11-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Bernicker, M.D., Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and materials on human subjects will be shared with other eligible investigators through appropriate means in accordance with the NIH policy on Sharing Research Data (NIH Guide, February 26, 2003). Data will be also shared with the funding agency and regulatory agencies as required. Data will be shared with other investigators within the limits of HIPAA and other patient confidentiality requirements. This will generally require removal of all patient identifiers for all source documents and the use of arbitrarily assigned one-way identifiers. In some cases, requestors will be asked to sign a formal data sharing agreement that will provide for a commitment to use data only for research purposes and not to identify individuals, keep the data secure, and destroy or return data after analyses are complete. Prior approval will be obtained from collaborating investigators, research sponsors, and/or other stake-holders before sharing if proprietary information or products are involved.
Supporting Information: Study Protocol

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was terminated early due to termination of funding by sponsor
Groups:
- Experimental: ADV/HSV-tk (5 x 1011 viral particles) in a 2-mL total volume will be injected intratumorally on day 0 of the study.
  Valacyclovir will be orally administered at a dose of 2 g three times daily for 14 days. Valacyclovir treatment will be administered 24 hours after the gene vector injection from day 1 to day 15 of the study.
  SBRT of 30 gray (Gy; 6 Gy X 5 fractions) will be administered over 2 weeks from day 2 to day 16 of the study.
  Nivolumab (480 mg) will be administered intravenously over 30 minutes every 4 weeks starting on day 17 of the study and continuing until disease progression, unacceptable toxicity, or up to 12 months in patients without disease progression.
  ADV/HSV-tk: Replication-defective recombinant adenovirus vector
  Valacyclovir: Prodrug of the antiviral drug acyclovir
  SBRT: Low-dose SBRT
  nivolumab: Fully human immunoglobulin (Ig) G4 anti-PD-1 monoclonal antibody
Period: Overall Study
Arm/Group | Experimental
Started | 11
Completed | 0
Not Completed | 11
Not completed — Physician Decision | 11

BASELINE CHARACTERISTICS:
Arm/Group | Experimental
Number analyzed (Participants) | 11
Age, Continuous [Mean (Full Range); unit: years] | 68.77 [59.54 to 85.25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Primary Diagnosis [Count of Participants; unit: Participants]
  Non-Small Cell Lung Carcinoma | 4
  Uveal Melanoma | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Determine the ORR of ADV/HSV-tk plus Valacyclovir therapy in combination with SBRT used as a window of opportunity treatment before nivolumab. Administration of ADV/HSV-tk + Valacyclovir in combination with SBRT before nivolumab represents a novel window of opportunity to enhance nivolumab efficacy by boosting endogenous immune-mediated antitumor activity and neoantigen expression.
  The concepts of the irRC are combined with RECIST 1.1 to come up with the modified irRC, which uses unidimensional measurements. For modified irRC, only target and measurable lesions are taken into account. The same assessment method and technique should be used to characterize each identified and reported target lesion(s) at baseline, during the trial, and at EOT. All measurements should be recorded in metric notation.
Time Frame: 30 days after the last dose of nivolumab, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 11
Participants
  Complete response (CR) | 0
  Partial response (PR) | 0
  Stable disease (SD) | 0
  Progressive disease (PD) | 11

2. Secondary Outcome: Overall Survival (OS) Rate
Description: Determine the OS rate. Months from start of treatment till date of death.
Time Frame: 30 days after the last dose of nivolumab, up to 6 months
Measure: Mean (Full Range); unit: Months
Arm/Group | Experimental
Number analyzed (Participants) | 11
Months | 15 [1 to 45]

3. Secondary Outcome: Progression Free Survival (PFS) Rate
Description: Determine the Progression Free Survival (PFS) rate.
  Progressive Disease (PD): At least a 20% increase in the sum of the diameters of target lesions, using the smallest sum on study (includes the baseline sum) as the reference. In addition to the relative 20% increase, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression)
  Overall irPD: ≥ 20% increase in the sum of the longest diameters of target and new measurable lesions increases (compared to nadir), confirmed by a repeat, consecutive observation at least 6 weeks (normally it should be done at 8 weeks) from the date first documented.
  Documentation of immune-related PD (based on modified irRC) does not mandate discontinuation of the study treatment even after irPD is confirmed with CT scan 6 weeks after the initial observation of irPD.
Time Frame: 30 days after the last dose of nivolumab, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 11
Participants | 0

4. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Estimate the CBR as assessed by RECIST 1.1 and modified immune-related criteria
Time Frame: 30 days after the last dose of nivolumab, up to 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental
Number analyzed (Participants) | 11
Participants
  Complete response (CR) | 0
  Partial response (PR) | 0
  Stable disease (SD) | 0
  Progressive disease (PD) | 11

ADVERSE EVENTS:
Time Frame: From informed consent signing up to and including 30 days after the last treatment dose of Nivolumab.
Arm/Group | Experimental
All-Cause Mortality (participants affected / at risk) | 1/11
Serious Adverse Events (participants affected / at risk) | 4/11
Other Adverse Events (participants affected / at risk) | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=11)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoglycemia (Blood and lymphatic system disorders) | 1 (1)
non-traumatic intracranial hematoma (Blood and lymphatic system disorders) | 1 (1)
Metabolic encephalopathy and dehydration (Metabolism and nutrition disorders) | 1 (1)
Progression of disease that resulted in Death (General disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental (N=11)
Weight loss (Metabolism and nutrition disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (General disorders) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Chills (General disorders) | 1 (3)
Constipation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Dehydration (General disorders) | 3 (3)
Bradycardia (Cardiac disorders) | 1 (1)
Confusion (Psychiatric disorders) | 3 (3)
Hyponatremia (Blood and lymphatic system disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthritic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cataract surgery (Eye disorders) | 1 (1)
Chest palpitations (Cardiac disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 6 (6)
Hypokalemia (General disorders) | 1 (1)
Inguinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intractable itchiness (General disorders) | 1 (1)
Loss of appetite (Metabolism and nutrition disorders) | 3 (3)
Migratory chest pain (Cardiac disorders) | 1 (1)
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Psoriasiform dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Night sweats (General disorders) | 1 (1)
Sleep disturbance (Nervous system disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Nasal discharge (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/33/NCT02831933/Prot_SAP_000.pdf